CLINICAL TRIAL: NCT04309799
Title: The Effect of Warm Compress Therapy Using the TearRestore Eyelid Warming Mask on Symptoms and Signs of Meibomian Gland Function
Brief Title: The Effect of Warm Compress Therapy Using the TearRestore Eyelid Warming Mask on Meibomian Gland Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-1960
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Dry eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single 10 minute session (Other): Study assessments will be performed before single 10 minute session of wearing the Tear Restore Mask and then study assessments will be repeated after the 10 minute single session has been completed.
  Interventions: Device: Tear Restore Mask
- Optional Extension (Other): Subjects can choose to extend use of the Tear Restore Mask at home for a period of 28 to 60 days. They will use the mask for a 10 minute time period one time per day and record the use in a diary.
  Interventions: Device: Tear Restore Mask

INTERVENTIONS:
Device: Tear Restore Mask — The Tear Restore Mask will be used for 10 minutes

SUMMARY:
This study plans to learn more about the effectiveness of the TearRestore eyelid warming mask on signs and symptoms of Meibomian Gland Dysfunction (MGD). MGD is a leading cause of dry eye symptoms. Warm compresses are a standard treatment recommended by physicians to treat those diagnosed with MGD. The study will investigate whether the TearRestore mask affects meibomian gland function and dry eye symptoms.

DETAILED DESCRIPTION:
The study will evaluate the effectiveness of the TearRestore eyelid warming mask on signs and symptoms of MGD. Warm compress treatments have been recommended as part of the standard of care by eye physicians, and are an important means in treating MGD. However, current treatment options suffer from varied temperature maintenance and poor compliance. The TearRestore™ mask offers patients a unique experience through providing sustained heat and the ability to see throughout the treatment, which will improve efficacy through improved compliance. If shown to be effective in altering Meibomian gland secretions at a single visit, this novel treatment could potentially offer the millions of patients suffering from MGD a more convenient and effective way to treat the condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (age 18-89) of any race, gender or ethnicity, diagnosed with meibomian gland dysfunction
* Symptom score greater than eight on the SPEED questionnaire
* Less than 75nm lipid layer thickness (LLT) utilizing the Lipiview II
* Less than 10 second tear break up time (average of 3 measurements)

Exclusion Criteria:

* Participants with less than 6/15 meibomian glands yielding liquid secretions in either eyelid
* Diagnosed with a systemic autoimmune condition including but not limited to Sjogren's or Lupus

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Standardized Patient Evaluation of Eye Dryness (SPEED) Questionnaire | Up to 60 days
  The SPEED questionnaire will be completed by the subject prior to using the Tear Restore Mask and then repeated after the 10 minute session

SECONDARY OUTCOMES:
Lipid Layer Thickness | Up to 60 days
  The Lipid Layer Thickness will be measured prior to using the Tear Restore Mask using the Lipiview II machine and then repeated following the 10 minute session.
Tear Breakup Time | Up to 60 days
  The Tear Breakup Time will be measured prior to using the Tear Restore Mask by the Clinician and then repeated following to 10 minute session.
Number of Meibomian Glands Yielding Liquid Secretions | Up to 60 days
  The Number of Meibomian Glands Yielding Liquid Secretions will be counted by the clinician prior to using the Tear Restore Mask and then recounted by the clinician following to 10 minute session.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hauswirth, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Dept. of Ophthalmology, Aurora, Colorado, United States